## 12/8/20

Title: Attitudes Towards Receiving Mental Health Care Using Telehealth During the COVID-19 Pandemic

NCT04693052

## Statistical Analysis

The most of the data was analyzed using SPSS(IBM Corp. Released 2020.) and Microsoft Excel(Microsoft Corporation) and some data was analyzed using R (R. Core Team, 2021; R. Studio Team, 2021). Descriptive statistics were calculated, which included number of participants and percentage of participants with a particular rating, mean ratings, standard deviation, standard error, standard Cohen's d(effect size). Inferential tests included 1 sample t-tests evaluating if scale means significantly deviate from the neutral "0" (which was in-person same as telepsychiatry for quality of care, perceived benefits, wait-times and missed appointment items and neutral ratings for telepsychiatry for comfort, satisfaction, and ease of use) . p<0.05 was considered statistically significant.